CLINICAL TRIAL: NCT02549950
Title: Efficiency and Efficacy of Peizo-Coticision in Reducing Orthodontic Treatment Time: Randomized Clinical Trial
Brief Title: Efficiency of Piezo-Corticision in Accelerating Orthodontic Tooth Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AL Yousef (Other)
Collaborators: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor-Investigator, AL Yousef, Sally K Al Yousef BDS; AEGD; GPR; MSc-Orthodontics, King Abdullah International Medical Research Center
Organization: King Abdullah International Medical Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC13/261/R
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Malocclusion, Angle Class I; Malocclusion; Angle Class II Division 1
Keywords: Accelerated orthodontic tooth movement (AOTM); Peizo-corticission
MeSH Terms: conditions — Malocclusion, Angle Class I; Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional OrthodonticTreatment (Active Comparator): Conventional orthodontic mechanics: canine and incisor retraction
  Interventions: Procedure: Conventional Orthodontic Mechanics
- Accelerated Tooth Movement (Experimental): Accelerated orthodontics: Peizo-Corticision Accelerated canine and Incisor retraction
  Interventions: Procedure: Peizocorticision

INTERVENTIONS:
Procedure: Peizocorticision — Peizocorticision a non invasive procedure used in/ to accelerate orthodontic tooth movement
  Other Names: AOTM Accelerated Orthodontic Tooth Movement
  Arms: Accelerated Tooth Movement
Procedure: Conventional Orthodontic Mechanics — Full Fixed Orthodontic Appliance with conventional orthodontic Mechanics
  Other Names: Conv Orth Mech
  Arms: Conventional OrthodonticTreatment

SUMMARY:
The purpose of this study is to provide evidence on the effectiveness, the efficiency and efficacy of Peizo-Corticission in accelerating orthodontic tooth movement and reducing orthodontic treatment time.

DETAILED DESCRIPTION:
1 Aim of the study- Part I:

This prospective controlled clinical trial (CCT), Split Mouth Design is conducted to assess the efficiency of piezo-corticision in accelerating tooth movement and in reducing treatment time during retraction of canine teeth in class II div 1 subjects.

Specific aim- Part I:

A- To compare rate of tooth retraction between piezo-corticised and the conventionally orthodontically moved canines

B- To compare length of treatment of both approaches.

2- Objectives of the Study Part II:

This prospective randomized controlled clinical trial (RCT) is designed to assess the efficiency of piezo-corticision in accelerating tooth movement and in reducing treatment time during retraction of anterior teeth in class II div 1 and class 1 bi-maxillary protrusive subjects.

Specific aim Part II:

1. To compare rate of tooth retraction between piezo-corticised and the conventionally orthodontically moved incisors
2. To compare length of treatment of both approaches.
3. To evaluate the quality of treatment outcome of both treatment approaches according to American Board of Orthodontics (ABO) standards.

ELIGIBILITY:
Study Subjects for Part I and Part II:

Inclusion:

* Voluntary participation of patients only
* Able to follow instruction, able to understand the consent form and sign it.
* Adult Female and Male Saudi patients 15-35 y.o
* Subjects who are none smokers
* Subjects with good health according to American Society of Anesthesiology ASA-I with full permanent dentition regardless of the third molars.
* Subjects with good periodontal and gingival health: Gingival Index GI≤ 1
* Subjects with a none gummy smile,
* Subjects with full complement of permanent caries-free dentition; Restored teeth should be of proper sound intact fillings
* Subjects without root anomalies
* Subjects with mild-moderate skeletal and dental cephalometric measurements: OB ≤ 40%, OJ ≤ 6, ANB ≤ 5 °, SN-GOGN ≤ 29 °, Subjects' dentition Angle classification class II div 1, 3mm molar and canine occlussal relationship; and subjects with class 1 Bi-maxillary protrusion

Exclusion:

* Subjects younger than 15 y.o
* Subjects who cannot comprehend the surgical procedure and who cannot consent for themselves
* Subjects who are medically classified as ASA-II, III
* Subjects who are taking any systemic or local medications especially Insulin, non-steroidal anti-inflammatory drugs, bisphosphonate, corticosteroids
* Subjects who are pregnant
* Subjects who are smokers
* Subjects with craniofacial syndromes: cleft lip and palate; or facial trauma
* Subjects with unhealthy or compromised periodontium
* Subjects with a gummy smile
* Subjects with inadequately treated endodontic and dental fillings problems
* Subjects with previous root resorption or dental developmental anomalies
* Subjects who had previous orthodontic treatment
* Subjects with TMJ signs and symptoms; Mandibular functional shift
* Subjects with extreme skeletal and dental class II: SN-GOGN ≥ 32°, OJ ≥ 6mm
* Subjects will be excluded if broken brackets or lost coils which have not been replaced immediately within few days from breakage or loss.
* Subjects will be excluded if any of mini-screws failed during treatment
* Subjects who become medically unfit during course of trial

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Rate of orthodontic canine movement | 4-6 months

SECONDARY OUTCOMES:
Rate of orthodontic Incisor Retraction | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sally K Al-Yousef, MSc-Ortho, Principal Investigator — KAIMRC
Locations (1):
- National Guard Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Mathews DP, Kokich VG. Accelerating tooth movement: the case against corticotomy-induced orthodontics. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):5-13. doi: 10.1016/j.ajodo.2013.04.008. No abstract available. PMID 23810039